CLINICAL TRIAL: NCT05900570
Title: The Effect of Acute Peri-Urethral Neurostimulation on Intra-Urethral Pressure In Women With Stress Urinary Incontinence (SUI) - Urodynamic Early Feasibility Study
Brief Title: Effect of Peri-Urethral Stimulation on Intra-Urethral Pressure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Corewell Health East (Other)
Responsible Party: Principal Investigator, Kenneth M Peters, MD, Director and Chair of the Department of Urology, Corewell Health East
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2023-117
Record Dates: First submitted 2023-05-13; First posted 2023-06-12 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Intervention Model Description: Participants who meet all eligibility criteria will be enrolled in the study and undergo urodynamic testing and LPP with and without neurostimulation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Urodynamic testing and LLP with and without pudendal nerve stimulation (Experimental): Commercially available stimulation needles or leads will be inserted into the peri-urethral space targeting the perineal branch of the pudendal nerve. An external neurostimulator settings will be adjusted to deliver acute stimulation. Urodynamic testing will be completed by filling the bladder to a set volume and observing for urinary leakage. The assessment will be completed with stimulation turned on and off. The neurostimulator device settings will be adjusted by the investigator to stay within safe and comfortable levels for each individual study participant.
  Interventions: Diagnostic Test: Urodynamic testing with and without pudendal nerve stimulation

INTERVENTIONS:
Diagnostic Test: Urodynamic testing with and without pudendal nerve stimulation — A urodynamic test with and without neurostimulation will be conducted. The external neurostimulator device settings will be adjusted to deliver acute nerve stimulation per the individual tolerance level to assess the effect on urethral pressure. A leak point pressure (LLP) during Valsalva maneuver will be assessed with and without acute nerve stimulation.

SUMMARY:
The purpose of this early feasibility prospective study is to gain initial understanding of the effect of acute peri-urethral neurostimulation on the perineal nerves on intra-urethral pressure.

DETAILED DESCRIPTION:
In this study intra-urethral pressure data will be collected and analyzed with and without peri-urethral neurostimulation. This is a single arm feasibility study of women diagnosed with stress urinary incontinence. The data collected may help researchers have a better understanding of the effect, if any, on neurostimulation on stress or mixed urinary incontinence. After informed consent and all eligibility criteria are met, enrolled participants will be brought in for a stimulation visit. At the stimulation visit, participants will undergo urodynamic testing with and without stimulation. A prophylactic antibiotic will be given before the procedure and a local anesthetic cream will be applied topically to the peri-urethral area. The participant will be prepped for urodynamic testing per protocol. Commercially available simulation needles or leads and external neurostimulator device will be used to perform peri-urethral neurostimulation of the perineal branch of the pudendal nerve. The amplitude will gradually be increased and intra-urethral pressure will be recorded. Stimulation parameters such as amplitude, pulse-width, and frequency will be explored to assess their effect on urethral pressure. Amplitude progressively will be increased until discomfort is noted, no further pressure increases are observed, or maximum output is achieved. When a consistent pressure is observed, record intra-urethral pressure measurements with stimulation on and off. Next, Leak Point Pressure (LPP) testing with and without stimulation will be completed. Start the urodynamic saline infusion until desired volume is reached. Observe for urinary leakage. This will be repeated with the stimulation on.

ELIGIBILITY:
Inclusion Criteria:

* Female aged 18 years old or older
* Capable of understanding the clinical study procedures and giving informed consent
* Willing and able to undergo the study procedure
* Diagnosis of SUI or stress predominant mixed incontinence, for at least 6 months
* Provided authorization to use and disclose information for research purposes

Exclusion Criteria:

* Predominant urge incontinence per patient report or medical record
* Active symptomatic uncontrolled bladder instability as determined by the investigator
* Regularly or intermittently used a urethral catheter
* Active bladder cancer (currently undergoing or scheduled to undergo treatment for bladder cancer).
* Previous radiation treatment in the pelvic floor
* History or symptoms of cystocele, enterocele or rectocele of grade 3 or 4. Per the medical record or as determined by the investigator
* Current infection (urethritis, cystitis or vaginitis) as determined by investigator.
* Active herpes genitalis
* Unevaluated hematuria
* Currently taking, or has taken within 4 weeks prior to the screening/baseline visit, pharmacological treatment for SUI (including but not limited to, alpha adrenergics, and tricyclic antidepressants)
* Severe or uncontrolled diabetes, (defined as being a diabetic with a hemoglobin A1c of ≥10%) per patient medical record.
* History of drug/alcohol abuse, mental dysfunction, or other factors limiting her ability to cooperate fully
* Pregnancy test with positive result during screening or women who are breastfeeding
* Women who are pregnant and/or have given birth in the previous 12 months
* Have implanted active neurostimulators, pacemakers, or defibrillators; neurostimulators which are passive or that can be briefly turned off for the stimulation procedure are acceptable
* Known systemic neurological dysfunctions
* Severe coagulation disorders
* Medically unstable at time of study and unsafe to undergo urodynamic testing (UDT) as determined by the investigator
* Presence of an artificial urinary sphincter
* Any medical condition (e.g. Multiple Sclerosis, spinal cord injury, mobility) or uncontrolled chronic disease (e.g. renal diseases that requires dialysis) that would interfere with the patient's ability to comply with the protocol and/or may affect the outcome of this study or safety of the subject as determined by the investigator

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Born female
Enrollment: 20 (Estimated)
Dates: Start 2024-02-26 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
The effect of acute peri-urethral neurostimulation on intra-urethral pressure. | At stimulation visit, 1 day
  Intra-urethral pressure (measured in cmH2O) will be recorded with stimulation on and off.

SECONDARY OUTCOMES:
Safety and tolerability will be assessed in relation to the incidence of adverse events occurring within one week of stimulation visit. | One week after completing the stimulation visit
  Safety and tolerability of peri-urethral stimulation will be assessed in related to the incidence of adverse events reported.
Valsalva leak point pressure (LLP) in response to acute peri-urethral neurostimulation compared to no stimulation | At stimulation visit, 1 day
  Leak point pressure (measured in cmH20) will be collected during neurostimulation and without neurostimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Peters, MD, Principal Investigator — Corewell Health William Beaumont University Hospital
Locations (1):
- Corewell Health William Beaumont University Hospital, Royal Oak, Michigan, United States